CLINICAL TRIAL: NCT03586622
Title: Home Monitoring of IBS Patients: Long Term Effect of Low FODMAP Diet With Re-introduction and Probiotic Treatment VSL#3 on IBS Symptoms and Gut Microbiota
Brief Title: One Year Home Monitoring and Treatment of IBS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Colitis-Crohn Foreningen (Other); Ferring Pharmaceuticals (Industry); Calpro AS (Other); Muusmann forlag (Unknown); Statens Serum Institut (Other); Genetic Analysis AS (Unknown)
Responsible Party: Principal Investigator, Pia Munkholm, MD and Professor in eHealth and epidemiology, Nordsjaellands Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H16023499
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: eHealth; Dietary Modification; Probiotics; Microbiome; Irritable Bowel Syndrome
Keywords: Home monitoring; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FODMAP diet (Experimental): Low FODMAP diet (LFD) Each IBS patient randomized to the Australian exclusion diet, Low FODMAP diet (LFD) group (n=52) will when allocated to LFD group have a one-hour counseling to the LFD by a nutritionist at the hospital. Within this one hour a diet anamnesis of the patient will be made in order to register the High FODMAP foods the patient is consuming (important that one find good low FODMAP substitutions). Based on the diet anamnesis optimization of the low FODMAP diet counseling can be made. They will receive hands-out with recipes, tips, meal plans, list of suitable low FODMAP foods and folder of foods they should avoid- most of information in the LFD folder patients will also find in the app 'Low FODMAP diet' which they will receive free of charge.
  Interventions: Dietary Supplement: Low FODMAP diet (LFD)
- VSL#3® (Experimental): Each IBS patient randomized to the probiotic VSL#3 arm (n=52) will at randomization be given VSL#3 for 4 weeks (56 sachets) together with a leaflet on VSL#3 - holding information on the product from the manufacture regarding storage, nutritional information etc. If the patients have any questions regarding the treatment, they can ask the project investigator handing out the VSL#3 to them. They will be instructed in taking their VSL#3 (2 sachets a day) as described by the manufacturer
  Interventions: Dietary Supplement: VSL#3®

INTERVENTIONS:
Dietary Supplement: Low FODMAP diet (LFD) — The Low FODMAP diet (LFD) is an acronym for Fermentable Oligo-, Di-, and Monosaccharides And Polyols - all of which are small osmotic active carbohydrates or sugar alcohols that are poorly absorbed in the small intestine and therefore easily fermented by the gut microbiota. The fact that they are fermented rapidly and osmotic active makes them potential and likely candidates for causing luminal distension due to accumulation of gas and water in the intestine.
  Arms: Low FODMAP diet
Dietary Supplement: VSL#3® — VSL#3® is a dietary supplement that helps maintain the balance of the intestinal flora. VSL#3® has been recognized and classified as GRAS (Generally Regarded as Safe) by a panel of experts in the USA for both adult and pediatric IBD and IBS patients. VSL#3® is a probiotic food containing 450 billion freeze-dried live lactic acid bacteria and bifidobacteria from 8 different strains per bag/sachet: Streptococcus thermophilus BT01, Bifidobacteria (B. breve BB02, B. longum* BL03, B. infantis* BI04), Lactobacillus acidophilus BA05, Lactobacillus plantarum BP06, Lactobacillus paracasei BP07, Lactobacillus delbrueckii subsp. bulgaricus** BD08; *Recently reclassified as B. animalis subsp. lactis ** Recently reclassified as L. helveticus. The recommended daily dose is 1-2 bags.
  Arms: VSL#3®

SUMMARY:
The purpose of this study Is to evaluate if a 4 weeks probiotic VSL#3 treatment and a strict LFD for 4 weeks are equally good in treating IBS symptoms in IBS patients with diarrhoea or mixed predominance and further evaluate the long term effect. Hopefully this one year individualized web-based IBS study will generate a fundament that could be used as a treatment in the primary care/sector to IBS patients.This one year study will be carried out based on an eHealth platform ibs.constant-care.com. Patients will self-measure on the web-program the first 4 weeks before randomization. The patients will fill out different questionnaires regarding symptom severity, adherence, stool consistency and frequency, quality of life, disease course type, food registration and weight. Nearly all of the questionnaires are illustrated to the patients in a traffic light manner (Green, Yellow and Red). They will also self-measure Fecal calprotectin on their smart phones and send in fecal samples for microbiome analysis. In this randomized cross over study - 104 IBS patients will be randomized to either a diet low in FODMAPs (fermentable, oligo-, di- and monosaccharides and polyols, LFD) or the probiotic product VSL#3® for 4 weeks. The probiotic group will receive 2 sachets a day (450 billions live bacteria in one sachet) for 4 weeks. After 4 weeks intervention (LFD or VSL#3) non responders, defined as a reduction of less than 50 points in IBS-SSS will after two weeks wash out period be crossed over. IBS patients randomized to LFD and responds to LFD will after a reintroduction counselling with dieticians at North Zealand university hospital after 4 weeks on a strict LFD start reintroducing high FODMAP foods until symptom flare (individual defined as either Yellow or Red, >175 in IBS-SSS). Hereafter they will go on a strict LFD again until symptom remission (IBS-SSS below 175, Green zone) - LFD responders will continue with this procedure for 10 months. IBS patients initially randomized to VSL#3 and are after 4 weeks of intervention characterized as responders will not be offered a LFD. Instead they will self- measure on the web with no intervention after the 4 weeks of VSL#3 treatment. When/if they reach a symptom flare ( again individually defined as either Yellow or Red, >175 point in IBS-SSS) they will be offered another 4 weeks VSL#3 treatment.

DETAILED DESCRIPTION:
IBS (irritable bowel syndrome) patients will be recruited from the out-patient clinic of North Zealand University Hospital, capitol region of Copenhagen, Denmark. Project investigator will give the patients all relevant information and forms needed to obtain a written informed consent. 104 IBS patients with diarrhoea or mixed type predominance will be included. Before enrollment, Patients will receive education on IBS and good toilet habit (squatty potty) etc. They will hereafter self-measure on a web-program the first 4 weeks in order to capture intra individual variation on the web and giving the patients time to learn how to use the 'tool': ibs.constant-care.com, in particular the primary end point IBS-SSS will be filled out several times during the first 4 weeks. The web algorithm for ibs.constant-care.com is specially designed for this trial. After 4 weeks on the 'web' IBS patients will be randomized to either Low FODMAP diet (LFD) or VSL#3 probiotic treatment (900 billions live bacteria/day) for 4 weeks. Patients randomized to the LFD group will be educated by a nutritionist in the diet and taught how to use a Danish Low FODMAP diet app in order to adhere to the LFD.

Non-responders (IBS-SSS<50) after 4 weeks intervention will have a 2 weeks wash out period and crossed over to the other intervention. LFD Responders (IBS-SSS ≥50) will be taught by a nutritionist at North Zealand University Hospital how to re-introduce foods high in FODMAPs and while re-introducing tightly monitor on the web-program. If LFD responders during the reintroduction period (10 months) will encounter a symptom flare individually defined as either Yellow or Red (that is > 175 on IBS-SSS) they will start on a strict LFD until symptom remission (<175 IBS-SSS) and so forth during the rest of the year. Responders to VSL#3 (IBS-SSS ≥50) will self-monitor on the 'web' and if the patients experience a symptom flare (again individually defined as either Yellow or Red - that is > 175 on IBS-SSS), they will be offered another 4 weeks VSL#3 treatment.

20 healthy controls will consecutively be included in the study and followed for a year on the web as well - they will not fill out as many questionnaires and is primarily included to have a background population and variation regarding the microbiome.

Patients will at inclusion receive their personal log in (Two Factor Authentication, 2FA) to ibs.constant-care.com and Calprosmart. Patients will register the below listed:

Severity scores system for IBS (IBS-SSS), web IBS-QoL (Quality of life), web Copenhagen IBS disease course, web Bristol Stool Chart and frequency, web FODMAP adherence rating scale (FARS), web Medication Adherence Rating Scale (MARS), web Evaluation questionnaire of the web program, web Evaluation questionnaire on food habits, web Fecal calprotectin (FC) on any smart Phone (CalproSmart app) Microbiome (patients will send in 2 fecal samples every time they send in samples - one for microbiome analysis (research biobank) and another one for a fecal biobank for future use. Weight, web IBS-SSS, QoL, BSC and frequency, FARS, MARS, FC, weight/BMI will be illustrated longitudinally to the patients in a traffic light manner (for ease of interpretation).

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the Rome III criteria for IBS.
* IBS patients classified as diarrhea or mixed type by the Bristol stool chart.
* Within normal BMI range (18.5-25)
* IBS patients who can read, speak and understand Danish
* Have a smart phone
* IBS patients that can manage going on Internet and wireless networks
* Above 18 years of age
* IBS-SSS>175

Exclusion Criteria:

* IBS Patients with diagnosed co-morbidities like diabetes
* IBS patients that have undergone gastrointestinal surgery
* IBS patients on IBS medication
* IBS patients on alternative diets
* IBS patients diagnosed with celiac disease and lactose intolerance
* IBS patients with severe mental disturbance or alcohol/ other drug abuse.
* IBS diagnosed with predominate constipation or unspecified
* Has previously been on low FODMAP diet (Guided by professional nutritionist )
* Has been on any probiotic or antibiotic treatment within 3 months prior to inclusion
* IBS patients with a BMI below 18.5 and above 25
* IBS patients with a language barrier
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-09-23 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Symptom Severity (5-Item visual analogue scale, IBS-SSS) | 4 weeks
  The IBS-SSS scale is constructed as a five item visual analog scale (VAS) which will be self-administrated by the patients on the web program. And results will be illustrated as a function of time in a traffic light manner to the patients (Mild, Green Zone <175, Moderate, Yellow Zone 175-300 and Severe, Red Zone > 300 on the IBS-SSS). IBS-SSS evaluates the intensity of IBS symptoms during the past 10 days with regards to: abdominal pain, distension, bowel habits, and interference with life in general. Each of the five items generates a maximum score of 100, which gives a maximum total score of 500 for all five items. A greater score indicates more severe symptoms. A cut off value for improvement/ responder of 50 point was recommended by Francis et al. 1997 and will also be used in this study to evaluate respond rates in the 2 arms.

SECONDARY OUTCOMES:
Symptom Severity (IBS-SSS) area under the curve (AUC) | 11 months
  The IBS-SSS scale is constructed as a five item visual analog scale (VAS) which will be self-administrated by the patients on the web program. Each of the five items generates a maximum score of 100, which gives a maximum total score of 500 for all five items. Results will be illustrated as a function of time in a traffic light manner to the patients (Mild, Green Zone <175, Moderate, Yellow Zone 175-300 and Severe, Red Zone > 300 on the IBS-SSS).
  The cumulative AUC for IBS-SSS, Red Zone, Yellow zone and Green zone after 11 months on the web program ibs.constant-care.com will be used for long term evaluation of the effect of the interventions.
Disease course, Copenhagen IBS Disease course Type | one year
  Based on epidemiology four figures have been developed to describe disease-course of IBS. These figures have been used in a retrospective study (Maagaard et al. 2016) to measure change in IBS disease course in IBS and IBD with co-existing IBS before and after a low FODMAP diet. The four figures depicting different types of disease courses is described as follows:
  1. Mild IBS with indolent course
  2. Mild IBS with aggressive course
  3. Chronic IBS with continuous course
  4. Chronic IBS with intermittent course The patients have to choose one figure representing their disease course type the best at inclusion and one year later.
Compliance, FODMAP adherence Report scale (FARS) | 4 weeks
  FODMAP Adherence Report Scale (FARS) was constructed to evaluate dietary adherence and was inspired by the validated Medication Adherence Report Scale by Byrne et al 2005. It consists of five questions regarding changing the diet, substituting the diet, forgetting to follow the diet and stop following the diet. Each of the five questions can be answered with the following options: 'always', 'often', 'sometimes', 'rare', and 'never' (scoring 1-5 points). A total score of 21 points or more (≥80%) will be considered as adherence to the diet (Maagaard et al. 2016).
Compliance, Medication Adherence Report Scale (MARS) | 4 weeks
  This questionnaire is measuring compliance to any medical/probiotic therapy by five questions with the following response options: always, often, sometimes, seldom, never (scoring 1-5 points). A total score of 21 points or more (≥80%) will be considered as compliant
Stool consistency, Bristol Stool Chart | 4 weeks
  To evaluate stool consistency, the Bristol Stool Scale will be used. The scale is composed of a simple visual chart accompanied by a text description that classifies stools in seven forms. The description differentiates among the following: type 1, separate hard lumps, like nuts; type 2, sausage-shaped but lumpy; type 3, like a sausage or snake but with cracks on its surface; type 4, like a sausage or snake, smooth and soft; type 5, soft blobs with clear-cut edges; type 6, fluffy pieces with ragged edges, a mushy stool; and type 7, watery, no solid pieces
Low grade inflammation measured by Fecal calprotectin (FC) on any smart phone | One year
  Calprotectin can be measured in stool and is a very sensitive marker for inflammation in the gastro intestinal tract. In IBS patients the use of this fecal biomarker is relative to patients with e.g. ulcerative colitis less clear but is used in this study for the purpose to detect low grade inflammation: below 200 mg/kg by using a FC home test, CalproSmart ((https://www.youtube.com/watch?v=wrTk7VumnSE).)
Microbiome | 4 weeks and one year
  The microbiome (same fecal samples) will be analyzed in 2 different ways.
  1. The method is based on culture independent 16S rRNA next generation sequencing. DNA from the patient fecal samples will be purified and 16S rRNA specific DNA will be amplified by polymerase chain reaction (PCR) technique of variable regions of the 16S rRNA gene and subsequently sequenced using Illumina 2x251 bp paired end sequencing on a MiSeq sequencing instrument.
  2. The dysbiosis index is based on polymerase chain reaction (PCR) technique of variable regions of 16S rRNA with selected 54 bacterial probes. Outcome from this analysis is a dysbiosis index (DI) ranging from 1 to 5 where 1 and 2 is defined as normobiotic and 3-5 is dysbiotic (5 more dysbiotic than 3 and 4). DI 'grade 1 and 2' is 'green' and defines normobiosis. Grade 3 I yellow and 4 and 5 is red (dysbiotic).
Symptom Severity (Time to and time in symptom remission, IBS-SSS) | 11 months
  The IBS-SSS scale is constructed as a five item visual analog scale (VAS) which will be self-administrated by the patients on the web program. Each of the five items generates a maximum score of 100, which gives a maximum total score of 500 for all five items. Results will be illustrated as a function of time in a traffic light manner to the patients (Mild, Green Zone <175, Moderate, Yellow Zone 175-300 and Severe, Red Zone > 300 on the IBS-SSS). Symptom remission is defined as green zone. We will count number of days (Survival curves ) that it takes for patients to reach green zone (symptom remission); less than 175 in IBS-SSS and time (days) in the green zone throughout 11 months.
Quality of life, IBS-QOL | Every 4 weeks
  The IBS-QoL is a self-report QoL measure.The IBS-QoL consists of 34 items, each with a five-point response scale: Items 1, 2, 4, 8-10, 12, 13, 16, 25-29, 34: answer options: 1 = not at all 2 = slightly 3 = moderately 4 = quite a bit 5 = extremely. And regarding the items 3, 5-7, 11, 14, 15, 17-24, 30-33 the answer options are : 1 = not at all 2 =slightly, 3 = moderately, 4 = quite a bit, 5 = a great deal. The 34 items are based on the following eight variables; dysphoria, interference with activity, body image, health worry, food avoidance, social reactions, sexual relationships.
  The individual responses to the 34 items are summed in a total score (max score 170) and the recall period is the past month (Patrick, D. L, 1998). The individual responses to the 34 items are summed up and averaged to give a total score and then transformed to a 0-100 scale for ease of interpretation with lower scores indicating better IBS specific QoL.
Food registration | Every 4 weeks
  Self-made food questionnaire consisting of 12 questions about food habits the last 4 weeks. Patients including Healthy controls fill it out on the web-app, Constant Care. The purpose of it is to capture any changes the last month that could worsen or improve IBS symptoms and therefore influence the effect of the two interventions: VSL#3 or the Low FODMAP diet. The questionnaire is constructed in such a manner that the patients answer on the web app in 12 text boxes and after filling out all text boxes the patients click the button 'send'. To each question and text box is a link to 'a good example' how to answer each question in regard to units, however, the patients can use any units they please.
Patients feedback for improvement of the ehealth platform | One year
  In order to improve the web program for future use. A self-made questionnaire has been made consisting of 11 question regarding the use of the web program Constant Care. Patients will fill out the questionnaire at follow up (that is after one year on the web program).
  The questionnaire consists of 9 binary questions e.g.: Did the project live up to your expectations? (Yes/No)
  Two additional questions were added:
  1. How long time have you used (average) when you have made registrations on the web app?
  2. List in the below text box any suggestions for improvements of the web app and click the button 'send'

CONTACTS AND LOCATIONS:
Overall Officials: Pia Munkholm, Professor, Study Director — North Zealands University Hospital
Locations (1):
- North Zealand university hospital, Gastro unit, Frederikssund, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ankersen DV, Weimers P, Bennedsen M, Haaber AB, Fjordside EL, Beber ME, Lieven C, Saboori S, Vad N, Rannem T, Marker D, Paridaens K, Frahm S, Jensen L, Rosager Hansen M, Burisch J, Munkholm P. Long-Term Effects of a Web-Based Low-FODMAP Diet Versus Probiotic Treatment for Irritable Bowel Syndrome, Including Shotgun Analyses of Microbiota: Randomized, Double-Crossover Clinical Trial. J Med Internet Res. 2021 Dec 14;23(12):e30291. doi: 10.2196/30291. PMID 34904950